CLINICAL TRIAL: NCT03716843
Title: Design of a Dynamic Pressure Monitoring System for Orthotic Treatment of Scoliosis
Brief Title: Dynamic Pressure Monitoring System for Orthotic Treatment of Scoliosis
Status: Recruiting | Type: Observational
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Washington University School of Medicine (Other); The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Joanne Yip, Professor, The Hong Kong Polytechnic University
Other Study IDs: GRF2019
Record Dates: First submitted 2018-10-20; First posted 2018-10-23 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Dynamic Pressure Monitoring

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pressure monitoring system for AIS: Adolescent idiopathic scoliosis (AIS) patients
  (1) all target subjects are aged 10 to 15 years old with immature skeletons (Risser grade 0-2); (2) they are diagnosed with AIS with a Cobb angle between 25-45° and high risk for curve progression; (3) the types of scoliosis are classified by the Lenke classification system; and (4) the subjects have received rigid brace treatment.
  Interventions: Other: Pressure monitoring system

INTERVENTIONS:
Other: Pressure monitoring system — The pressure measurement undergarment will be given to all consenting AIS patients who have received their own thoraco-lumbo-sacral orthosis (TLSO) rigid brace. Each patient will wear the undergarment first and the TLSO brace on top. FBG sensors embedded in the undergarment will measure each pressure signal at approximately 2 minutes. The average force reading will be calculated.
  Then, the experiment will be repeated once, but the anisotropic textile brace will replace the TLSO brace. The pressure measurement system will be used to obtain an accurate and adequate comparison of the forces applied to the patients. The effectiveness of the anisotropic textile brace will be evaluated through X-ray radiography, and its correction effect with be compared with that of the TLSO brace.
  Other Names: Pressure measurement undergarment

SUMMARY:
Adolescent idiopathic scoliosis (AIS) involves three-dimensional spinal deformity in children aged between 10 and 16. Traditional braces modify the natural dynamics and thus the mechanical behaviour of the scoliotic spine through external constraints. Patients usually develop pressure ulcers and skin irritation when prescribed brace treatment for 18-23 hours per day. The excessive pressure, unknown pressure distribution and pressure shifting between the human body and the brace causes the effects of brace treatment to be unpredictable. Dynamic pressure monitoring system will be developed based on the body landmarks of scoliotic patients and critical areas where active pressure is applied by the brace. The overall pressure distribution and dynamic pressure between the body and the thoraco-lumbo-sacral orthosis (TLSO) rigid brace will be measured. The efficacy of the brace design will be evaluated, and the maximum compressive stresses that patients can endure on different body parts without pressure injury can be computed.

DETAILED DESCRIPTION:
Global rates of adolescent idiopathic scoliosis (AIS) range from 0.9% to 12%, and within this population, approximately 10% of adolescents aged 10-16 will eventually need treatment. The most common conservative treatment is bracing, in which AIS patients are prescribed a brace for 18 to 23 hours daily until skeletally mature. The objective of bracing is to stop curve progression and restore normal alignment of the spine by active pressure from the brace. There is strong clinical evidence of a positive correlation between the tightness of daily brace application and the ability of the brace to decrease the risk of curve progression to a surgical threshold. However, patients suffer physical and functional discomfort resulting from pressure points, including pressure ulcers, skin irritation and even asthma attacks, which reduces compliance with brace treatment. Clearly, the knowledge of human body responses to pressure applied by brace treatment remains lacking.

This multi-disciplinary collaborative study involves experts in electrical and electronic engineering, orthopaedics, materials science and textiles, and biomechanics. A revolutionary pressure measurement system that integrates fibre optic sensors with textile yarns will be developed in the form of an undergarment. The sensor arrangement in the undergarment will be designed according to the body landmarks of scoliotic patients and critical areas where active pressure is applied by the brace. The overall pressure distribution and dynamic pressure between the body and the scoliosis brace will be measured. The efficacy of the brace design will be evaluated, and the maximum compressive stresses that patients can endure on different body parts without pressure injury can be computed.

Academia, clinicians and AIS patients are predicted to benefit from using the pressure system, which determines the optimum pressure to be exerted on patients while minimizing pressure injuries. The output of the project can be extended to the standardization of pressure levels applied by different orthotic devices and will add a new dimension to fibre optic applications in biomechanics.

ELIGIBILITY:
Inclusion Criteria:

* Teenagers diagnosed with adolescent idiopathic scoliosis
* Cobb's angle between 25 to 45 degrees
* Immature skeletons (Risser grade 0-2)
* Types of scoliosis are classified by the Lenke classification system
* Have received rigid brace treatment

Exclusion Criteria:

* Contraindications for x-ray exposure
* Diagnosis of other musculoskeletal or developmental illness that might be responsible for the spinal curvature
* History of previous surgical treatment for AIS
* Contraindications for pulmonary and/ or exercise tests
* Psychiatric disorders
* Recent trauma
* Recent traumatic (emotional) event

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study will be divided into two phases. In Phase 1, an exploratory pilot study will be performed with up to two different braces tried on the same patient in one spinal centre in Hong Kong.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-01-02 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall pressure distribution and dynamic pressure | 2 hours after wearing the brace
  1. Dynamic Pressure Changes (kPa) Monitored Over 2 Hours of Brace Wear, as Measured by the Optical Fibre Sensors.
  2. Overall Pressure Distribution (kPa) Monitored Over 2 Hours of Brace, as Measured by the Optical Fibre Sensors.

SECONDARY OUTCOMES:
Scoliosis Research Society Quality of Life Questionnaire | 6 months after wearing the brace
  1. Change in Scoliosis Research Society Score (SRS-22r) for Quality of Life Before and After Brace Usage. It includes five domains that evaluate function, pain, self-image, psychosocial status and satisfaction with the treatment and will be distributed to both experimental and control groups at 0 and 6 months. It has a minimum score of 22 and a maximum score of 110, with higher scores representing greater patient quality of life.
Visual analogue scale | 6 months after wearing the brace
  1. Change in Visual Analogue Scale (VAS) Scores for Pain Before and After Brace Usage.
  VAS is a straight horizontal line measuring 100 mm. The ends are defined as the extreme limits of pain, oriented from the left at 0 mm to the right at 100 mm. Typically, higher scores indicate a worse outcome, i.e., more pain.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Yip, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Tsim Sha Tsui, Kolwoon, Hong Kong

IPD SHARING:
Plan to Share IPD: No